# The effects of a personalized sleep improvement App from SleepScore Labs: a single-blinded randomized waitlist controlled trial

| Title | The effects of a personalized sleep improvement App from SleepScore Labs: a single-blinded randomized waitlist controlled trial |
|---|---|
| Protocol version identifier | Apr 28, 2023 (replaces previous version from Jan 26, 2023) |
| Product | SleepScore Labs App commercially distributed for measuring sleep and providing sleep advice based on a dynamic and personalized advice engine. |
| Sponsor | ResMed Germany Inc., Fraunhoferstr. 16, 82152<br>Martinsried, Germany |
| Research question and | Primary objective: |
| objectives | To assess changes in subjective sleep quality measured using validated questionnaires (SF-B) between active sleep-improvement condition through the Dein Schlaf. Dein Tag. App and waitlist condition after 6 weeks and 12 weeks Secondary chiestings. |
| | <ul> <li>Secondary objectives: <ul> <li>To assess changes in further metrics between app condition and waitlist condition comparing baseline with 6 weeks and 12 weeks follow-up including feeling of being refreshed in the morning, overall sleep complaints, and health measures using validated questionnaires (PSQI, PSS, SF-12, SF-B). Within the app condition, six objective sleep parameters (sleep onset latency, wake after sleep onset, total sleep time, sleep efficiency, sleep staging, nighttime awakenings) will be assessed by comparing baseline with 6 weeks and 12 weeks follow-up.</li> </ul> </li> </ul> |
| Country of study | Germany |
| Author | <ul> <li>Christoph Schöbel (Principal Investigator)</li> <li>Elie Gottlieb (Primary SSL)</li> <li>Daniela Ehrsam-Tosi (Primary ResMed)</li> <li>Susanne Fischer (Secondary ResMed)</li> </ul> |

# Marketing authorisation holder(s)

| Legal representative in Europe: ResMed Germany Inc.,<br>Fraunhoferstr. 16, 82152 Martinsried, Germany |
|---|
| Phone: +49 (0) 89 99 01-001<br>Fax: +49 (0) 89 99 01-10 08 |

# 1. Table of contents

| 1. | Table of | contents | 3 |
|----|-----------|---------------------------------------------------|----|
| 2. | List of a | bbreviations | 5 |
| | 2.1 De | claration of Helsinki and Signatures | 6 |
| 3. | Abstract | <u> </u> | 7 |
| 4. | Amendr | nents and updates | 9 |
| 5. | Milestor | nes | 10 |
| 6. | Rationa | le and background | 11 |
| 7. | Researc | ch question and objectives | 12 |
| 8. | Intensity | of Use | 12 |
| 9. | Researc | ch methods | 12 |
| | 9.1 Stu | udy design | 12 |
| | 9.2 Ra | ndomization and allocation concealment | 13 |
| | 9.3 Bli | nding | 13 |
| | 9.4 Ty | pe/Design of study | 13 |
| | 9.4.1 | CONSORT Study Flow Diagram | 14 |
| | 9.4.2 | Primary Endpoint | 14 |
| | 9.4.3 | Secondary Endpoints | 15 |
| | 9.4.4 | Study population | 15 |
| | 9.4.5 | Study duration | 16 |
| | 9.4.6 | Withdrawal from the trial | 16 |
| | 9.4.7 | Compensation | 16 |
| | 9.4.8 | Sleep Measurement | 16 |
| | 9.4.9 | Intervention and Control | 16 |
| | 9.4.10 | Inclusion of users and baseline parameters | 17 |
| | 9.4.11 | Assessments Table | 18 |
| | 9.5 Da | ta sources | 18 |
| | 9.5.1 | Data obtained from users | 18 |
| | 9.5.2 | Data imported from the Dein Schlaf. Dein Tag. App | 18 |
| | 9.6 Stu | udy size | 18 |
| | 9.7 Da | ta management | 19 |
| | 9.7.1 | Personal data and data protection | 19 |
| | 9.8 Da | ta analysis | 20 |
| | 9.9 Qu | ality control | 20 |
| | 9.9.1 | Access to Source Data/Document | 20 |
| | 9.9.2 | Quality assurance: | 21 |
| | 9.10 Stu | udy monitoring | 21 |
| | 9.10.1 | Audit | 21 |

| 9.11 Limitations of the research methods | 21 |
|------------------------------------------------------------------|----|
| 9.12 Other aspects | 21 |
| 10. Protection of human subjects | 21 |
| 11. Management and reporting of Adverse Events/Adverse Reactions | 22 |
| 12. Plans for disseminating and communicating study results | 22 |
| Annex 1. Questionnaires | 22 |
| Annex 2 References | 22 |

# 2. List of abbreviations

| Abbreviation | Definition |
|---|---|
| GCP | Good Clinical Practice |
| GDPR | The General Data Protection Regulation |
| ICH-GCP | International Conference on Harmonisation on Good Clinical Practice |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| PSQI | Pittsburgh Sleep Quality Index |
| PSS | Perceived Stress Scale |
| SF-12 | Short Form 12 Health Survey Questionnaire |
| SF-B | Schlaffragebogen B |
| SOP | Standard Operating Procedure |

# 2.1 Declaration of Helsinki and Signatures

The undersigned have read this protocol and agreed to conduct this study in accordance with all stipulations of the protocol and in accordance with the Declaration of Helsinki.

| Date | Name and Signature |
|---|---|
| | Elie Gottlieb (Applied Sleep Scientist, SleepScore Labs) |
| | Daniela Ehrsam-Tosi Daniela Ehrsam-Tosi Daniela Ehrsam-Tosi (Director Medical Affairs CRS, ResMed) |
| | Susanne Fischer (Senior Manager Medical Affairs CRS, ResMed) |
| | Christoph Schöbel (UnivProf. Dr. med., Principal Investigator) |

| 2.1 | Declaration | of Helsinki | and Signatures |
|-----|-------------|-------------|----------------|
|-----|-------------|-------------|----------------|

The undersigned have read this protocol and agreed to conduct this study in accordance with all stipulations of the protocol and in accordance with the Declaration of Helsinki.

| Date | Name and Signature |
|------------|----------------------------------------------------------------|
| | Elie Gottlieb (Applied Sleep Scientist, SleepScore Labs) |
| | Daniela Ehrsam-Tosi (Director Medical Affairs CRS, ResMed) |
| | Susanne Fischer (Senior Manager Medical Affairs CRS, ResMed) |
| 09-05-2023 | Christoph Schöbel (UnivProf. Dr. med., Principal Investigator) |

# 3. Abstract

| Title | The effects of a personalized sleep improvement App from SleepScore Labs: a single-blinded randomized waitlist controlled trial |
|---|---|
| Rationale and<br>Background | The Dein Schlaf. Dein Tag. sleep improvement App powered by SleepScore has not yet been empirically validated in the long-term assessment and management of people in the general population suffering from sleep complaints but did not yet fulfill the clinical criteria of an insomnia disorder. |
| Research | Primary objective: |
| objectives | Assessed at baseline, 6 weeks and 12 weeks, improvements in self-reported sleep quality while using a dynamic and personalized sleep advice engine app will be compared to a waitlist control group. Secondary objectives: |
| | Assessed at baseline, 6 weeks and 12 weeks, improvements in mental health, sleep problems, and stress will be compared to a waitlist control group. In the intervention (app) group, changes in objectively measured sleep parameters (sleep onset latency, wake after sleep onset, total sleep time, sleep staging, nighttime awakenings) over 6 and 12 weeks will be studied. |
| Study design | Single-blinded randomized waitlist controlled trial |
| Population | Inclusion criteria: iOS user, or user of one of the following: Samsung Galaxy S7 Edge and S7, S8, S8+, S9, S9+, S20, S20 FE, S20+, S21 Ultra Samsung Galaxy Note 8 and 9 Regensburg Insomnia Scale (subclinical insomnia: Score 13-24) ≥ 18 years old. Naive to the SleepScore Labs App Able to fully understand information on data protection and provide written informed consent Not included in other treatments targeting sleep Exclusion criteria: Clinically significant sleep disorders (e.g. Restless legs disorders, sleep-related breathing disorders, parasomnias) Bedtime less than 6 hours Any of the following medical problems: |

| | <ul> <li>Current mental disorder affecting sleep (e.g., depression, anxiety disorders, bipolar disorder, schizophrenia)</li> <li>Current severe medical conditions (e.g. chronic pain, cancer)</li> <li>Any of the following medications/substance use: <ul> <li>Prescription of sleep medication or overthe-counter sleep medication (e.g., melatonin, "Hoggar night")</li> <li>Medication for other conditions (e.g., anxiety, ADHD) that affect sleep, e.g., antidepressants, antipsychotics.</li> <li>Consumption of 3+ units of alcohol on 4 or more nights per week</li> <li>Recreational drug use</li> </ul> </li> <li>Pregnant or nursing mothers</li> <li>Infant or child under age 1 at home</li> <li>Shift work</li> <li>Current use of other Sleep Tracking App's</li> </ul> |
|---|---|
| Variables | Questionnaire data will be collected at baseline, after 6 and 12 weeks. Objective sleep data will be collected using the SleepScore App, and stored within the Microsoft Azure cloud system, an ISO 27001 certified and SOC 1 and SOC 2 compliant cloud service provider. Self-reported questionnaire data will be captured using an EU data center of Forsta/Decipher which is GDPR compliant, ISO 27001 certified, with SOC2 accredited data centers. |
| Data sources | Data obtained from users: Baseline, 6-weeks, and 12-weeks measurements derived from validated questionnaires Data imported from the Dein Schlaf. Dein Tag. App: Objective sleep data, daily logging, and usage monitoring data recorded by the Dein Schlaf. Dein Tag. App |
| Study size | Overall, 600 users (300 app condition, 300 waitlist control group) will be included in Germany. |
| Data analysis | The questionnaire date will be analyzed by an ANOVA, with one factor (app condition vs. waiting list control group) and time (Baseline, 6-weeks, 12-weeks). To handle missing values, a mixed-model approach with the same factors will be applied. The |

critical statistical test would be the interaction term between app condition and the waiting-list control group. Objectively measured data will be analyzed using multi-level modeling (MLM) in a nested way (nights within participants), allowing for analyzing changes within the intervention (app) group. To evaluate changes in primary and secondary outcome measures assessed by validated scales at baseline, 6-weeks, and 12-weeks, we will compare within-group differences for each time-point using a t-test if normally distributed, or the Mann Whitney-U test for non-normally distributed continuous data. In addition, effect sizes for the changes within both groups (questionnaire data) and app group (objective sleep parameters) will be computed.

### 4. Amendments and updates

Amendment No. 1, Jan 26 2023 Amendment No. 2, Apr 28 2023

| Section | Amendment or update detail | Reason |
|---|---|---|
| 5 Milestones | Dates changed | Adapted according to preparation of study |
| 9.4 Design | Deleted "written", added "A participant information document with consent form will be provided with page-turning function. Participant has to agree that his/her data will be used in this study by clicking "yes, I agree" or "no I don't agree and do not want to participate"." | Electronic consent ensures a that participants can follow a defined workflow and pathway and will be guided smoothly through the recruitment portal. This avoids that too many potential participants are being lost during the course of recruitment. |
| 9.4.1 | Adapted flowchart: Informed Consent – then baseline assessment – then randomization | Now follows the routine in study practice. Before the randomization should have occurred before the baseline assessment. Since randomization means access to the app for the "app group", the timepoint of filling out the baseline questionnaire could have been after first app usage. This will be avoided when doing baseline before randomization and app download. |
| 9.5.1 Data | Deleted Munich Chronotype<br>Questionnaire | Conversion into electronic format problematic; would have compromised the outcomes |

| 9.5.1 Data | Deleted Landecker Inventar zur<br>Erfassung von Schlafstörungen<br>(LISST) | Study flow and assessment of participants for eligibility in the e-portal required a combination of in-/exclusion criteria with the LISST to ensure all screening criteria could be met. LISST is not required to be applied as a separate questionnaire. |
|---|---|---|
| 9.7.1 Data management | Deleted [], forwarded to SleepScore, there combined with objectively measured sleep data, and then securely shared with ResMed where it will be stored for 10 years." Added: "Objective sleep data from the app as collected and controlled by SleepScore Labs and self-reported questionnaire data as collected by a vendor on behalf of ResMed Objective sleep data from the Dein Schlaf. Dein Tag. App as specified in this protocol, and without personal identifiers will be send to vendor, combined with self-reported questionnaire data by vendor and equipped with new identifiers to result in a deidentified set of study data. []shared with Sleepscore Labs for joint analysis." Added: "Deidentified study data will be stored at ResMed for 10 years." | Changes were necessary to be compliant with EU-GDPR. Processes had to be restructured to prevent ResMed from potentially getting access to personal data of study participants. |
| Annex 1 | Deleted LISST | Not required as separate questionnaire. Accurate recruitment of participants through automated electronic assessment made a fusion of eligibility criteria necessary. |
| Annex 1 | Deleted Munich Chrontype<br>Questionnaire | Conversion into electronic format problematic; would have compromised the outcomes |
| Inclusion criteria | Added "Samsung Galaxy S7 Edge<br>and S7, S8, S8+, S9, S9+, S20,<br>S20 FE, S20+, S21 Ultra Samsung<br>Galaxy Note 8 and 9" | Increasing the number of active users of the application by also allowing other devices which have been validated to deliver a similar performance in running the app. |

# 5. Milestones

| Milestone | Planned date |
|--------------------|--------------------------------|
| Start of enrolment | January 2023 (actual) |
| End of enrolment | May 2023 (anticipated) |
| Final results | July/August 2023 (anticipated) |

#### 6. Rationale and background

Sleep disturbances have a documented impact on general mental and physical well-being across many domains (e.g., Cappuccio et al., 2010; Dinges et al., 1997; Knutson et al., 2007). It has been estimated that approximately 20-35% of individuals report moderate symptoms of poor sleep (Hillman and Lack, 2013). Sleep-wake dysfunction contributes to the pathogenesis and evolution of neuropsychiatric conditions including depression, anxiety, and chronic pain, and are associated with an increased risk of chronic neurological health conditions including cerebrovascular disease, cardiovascular disease and neurodegenerative disorders. Those with poor sleep may experience general dissatisfaction with sleep quality or quantity which may be associated with minor to moderate difficulty initiating or maintaining adequate sleep (Benca et al., 2005).

The cause of sleep-wake dysfunction may be attributed to a myriad of environmental (e.g., excessive bright light before sleep), cognitive (e.g., pre-sleep worrying and anxiety), behavioral (e.g., caffeine or alcohol consumption prior to sleep), and physiological factors (e.g., pre-sleep arousal). A variety of sleep improvement options exist for poor sleep including pharmacological interventions, over-the-counter sleep aids, and cognitive and behavioral interventions. While the preferred treatment for those with clinical threshold poor sleep is cognitive behavioral therapy for insomnia (CBT-i) delivered in person, this effective approach is both time-consuming and costly, with implementation limited by an unmet need for trained providers (Espie et al., 2001). Furthermore, studies suggest that many individuals with sleep difficulties do not seek professional help and report a preference for non-pharmacological and personalized, self-help strategies (Vincent and Lionber, 2001, Morin et al., 2006). Despite this, few evidenced-based sleep improvement digital programs exist founded on the principles of behavioral change psychology and sleep hygiene targeting non-clinical populations for primary prevention.

Due to poor sleep's multitude of causes (e.g., environmental, cognitive, behavioral, or physiological) and symptoms (e.g., long sleep onset latency, short sleep duration, elevated wake after sleep onset and nighttime awakenings, poor sleep quality), a personalized and dynamic sleep improvement program tailored to a user's lifestyle and specific needs may be required to help nudge users towards sleep-promoting behaviors and attitudes. Digital and mobile health platforms are also highly scalable and cost-effective, thus allowing for widespread implementation across larger populations.

The purpose of the present study is to conduct a randomized controlled trial to evaluate a digital smartphone application, the Dein Schlaf. Dein Tag. application powered by SleepScore, designed to improve sleep and sleep-permissive behaviors. The Dein Schlaf. Dein Tag smartphone application utilizes a dynamic and personalized sleep advice engine founded in the principles of behavior change psychology and sleep hygiene that offers a novel, non-invasive and non-pharmacological solution designed to improve sleep

outcomes in those with common sleeping difficulties. While the sleep measurement technology behind Dein Schlaf. Dein Tag. has already been previously validated against gold-standard polysomnography (Zaffaroni et al., 2019), its sleep improvement features have not yet been empirically validated in the long-term assessment and management of people in the general population with a broader range of sleep problems.

#### 7. Research question and objectives

The primary objective of the present study is to examine improvement regarding self-reported sleep quality when using the Dein Schlaf. Dein Tag. sleep improvement engine App when compared to a waitlist condition. Validated questionnaires will be administered to assess self-reported sleep quality, health perception, psychosocial factors and sleep-permissive behaviors (i.e., preventative health).

Due to the dynamic and personalized nature of the intervention and its potential impact on various sleep-wake parameters depending on the user's objectively measured sleep (only app condition) and self-assessed goals, we have chosen multiple secondary endpoints: sleep onset latency, wake after sleep onset and total sleep time will be used to determine sleep changes.

Participants will be required to complete the following tasks during the study period:

- 1. Start the sleep tracking device via a smartphone app before lying down in bed and turning off the lights to go to sleep (only for intervention (app) group).
- 2. In the morning, turn off the sleep tracking device as soon as they wake up and decide to leave the bed (only for intervention (app) group).
- 3. Log day and regularly use the different modules addressing different aspects of sleep, including advice for change (only for intervention (app) group).
- 4. At the three time points shown in 8.4.1 flow diagram, complete a longer questionnaire using an E-Link. These questionnaires will cover demographic information, subjective mental and physical health, subjective sleep, and stress level. (valid for app condition and waitlist control group)

#### 8. Intensity of Use

Although app condition participants will be instructed to track sleep and engage with the app every night, the minimal internal compliance threshold for intensity of use is set at 3 nights of tracking per week. If participants track less than 3 nights per week, they will receive up to 3 reminder follow-up emails. The primary analysis will include all randomized participants. Secondary analyses will be conducted using an adherent to treatment approach, excluding participants who did not sufficiently engage with app throughout the study (<3 tracked nights of sleep per week).

#### 9. Research methods

#### 9.1 Study design

The study is a randomized waitlist controlled trial of a sleep improvement app. The present study design is summarized in Figure 1. We decided to use a between-group design as we want to determine the effect of the sleep improvement app vs. not using anything, as the study app is aiming to improve subjective sleep quality in order to prevent progression to clinical relevant sleep problems (primary prevention). Participants will be randomly assigned to the Sleep Improvement App intervention or the waitlist condition. Online assessments will take place at Baseline (0 weeks), 6 weeks (during the intervention), and 12 weeks (after intervention).

#### 9.2 Randomization and allocation concealment

This study will use simple randomization with an allocation ratio of 1:1, as recommended for large randomized controlled trials. Randomization will be conducted by an automated online system; hence the research team will be unable to influence randomization and have no access to future allocations.

#### 9.3 Blinding

Assessments will be self-reported and carried out online, and the research team will be blinded to outcomes during the trial. Participants will be informed of their randomization outcome by an automatic email, and hence they will not be blinded to treatment allocation. It is notable that the study sponsors will not have any contact with research participants and will therefore be unable to bias the allocation or assessments. If participants do contact the team and reveal the allocation, the absence of assessments carried out by an investigator prevents any biases.

#### 9.4 Type/Design of study

Naïve participants will be consecutively enrolled into the trial and randomized into either the wait-list condition or Sleep Improvement App-condition, provided that all inclusion and exclusion criteria are met and consent is given to use their data according to data privacy regulations. A participant information document with consent form will be provided with page-turning function. Participant has to agree that his/her data will be used in this study by clicking "yes, I agree" or "no I don't agree and do not want to participate". Eligible participants will receive written information about all relevant aspects of the study and that their participation in the study is voluntary and they have the right to refuse or withdraw their consent at any time without negative consequences. The study has been registered with ClinicalTrials.gov (210915DSDT). This paper contains modifications, which will be submitted to the Ethics Committee for approval prior to implementation. The current and further amendments will be documented in detail in the ClinicalTrials.gov registry. On the consent form, participants will be asked if they agree to the use of their data in case of withdrawing from the trial. Participants will also be asked for permission for the research team to share relevant data with people from SleepScoreLabs and ResMed taking part in the research or from regulatory authorities, where relevant. This trial does not involve collecting biological specimens for storage.





#### 9.4.2 Primary Endpoint

Statistically significant improvement in subjective sleep quality measured using a validated questionnaire between active sleep-improvement condition through the Dein Schlaf. Dein Tag. App and the waitlist condition comparing baseline with 6 weeks and 12 weeks measures.

Self-report sleep parameters: Sleep Quality score (SQ) of the SF-B (9 Items)

#### 9.4.3 Secondary Endpoints

Improvements in sleep metrics between app condition and waitlist condition comparing baseline with 6 weeks and 12 weeks measures

Note, given the dynamic and personalized nature of the intervention and its potential impact on various self-assessed goals, we have chosen multiple secondary endpoints that we expect to see statistically significant sleep improvements in depending on baseline self-reported sleep parameters, including the following:

- Health measures including overall sleep problems, feeling of being refreshed in the morning, mental health stress (PSQI, PSS, SF-12, SF-B)
- Objective sleep parameters (only app condition): Total sleep time, sleep onset latency, wake after sleep onset, sleep efficiency.
- Self-reported app-based items in app condition group.

#### 9.4.4 Study population

This research aims to target a non-clinical population with sublinical sleep disturbances that is interested in improving their sleep. To ensure we recruit a non-clinical sample, we will exclude users who have indicated they have a diagnosed sleep disorder as well as those identified as being at high risk of a sleep disorder based on validated screening tools. This research has no specific recruitment goals with respect to race or ethnicity and will not base participant eligibility on such criteria. However, this information may be recorded as part of the data collected.

#### Inclusion criteria:

- iOS user, or user of one of the following: Samsung Galaxy S7 Edge and S7, S8, S8+, S9, S9+, S20, S20 FE, S20+, S21 Ultra Samsung Galaxy Note 8 and 9
- Regensburg Insomnia Scale (poor sleep indicated by a score of 13-24, excluding those without sleep problems and those with probable insomnia disorder)
- ≥ 18 years old.
- Naive to the SleepScore Labs App
- Not included in other treatments around sleep
- Able to fully understand information on data protection and provide written informed consent

#### Exclusion criteria:

- Bedtime less than 6 hours
- Any of the following medical problems:
  - Untreated psychological disorder affecting sleep (e.g., depression, anxiety disorders, bipolar disorder, schizophrenia)
  - Current severe medical conditions (e.g. chronic pain, cancer)
- Any of the following medications/substance use:
  - Prescription sleep medication or regular use of over-the-counter sleep medication
  - Medication for other conditions (e.g., anxiety, ADHD) that affect sleep, e.g. antidepressants, antipsychotics
- Consumption of 3+ units of alcohol on 4 or more nights per week
- Recreational or nightly drug use
- Pregnant or nursing mothers
- Shift work
- Travel across 2 or more time zones during study period
- Sleeping more than 7 nights not at home during study period
- Users who newly received a diagnosis of a sleep disorders
- Users who start sleep or other psychoactive medication during the study period

Use of other Sleep Tracking App's during the study period

#### 9.4.5 Study duration

Recruitment for the study will be rolling, Baseline Assessment is at week 0. A follow up is scheduled after 6 weeks and 12 weeks of both the app and waitlist group. The end of data collection is planned after 12 weeks from baseline of the last user included. Final intention to treat analysis of study data will subsequently be performed.

#### 9.4.6 Withdrawal from the trial

Participants are free to withdraw from the trial at any time without giving any reasons. They will not have any negative consequences in the relationship to SleepScore Labs or ResMed. In the event that a user withdraws consent, the date and reason for termination – if provided – will be documented. For participants who drop out of the study, assessments that are part of the study design will be conducted only if the participants agree.

#### 9.4.7 Compensation

All enrolled participants will receive 20 euros for completing each follow-up assessment including baseline, 6-weeks, and 12-weeks, paid at the end of the study. Regular use of the sleep app will be compensated with 50 Euros.

#### 9.4.8 Sleep Measurement

The Dein Schlaf. Dein Tag. application powered by SleepScore includes a polysomnography-validated non-contact sleep monitoring technology employing inaudible sonar to monitor the movements and respiration of a participant in bed. A validation study of the sonar technology against gold-standard polysomnography showed high sensitivity (88%) and specificity (65%), exceeding agreement that is typically reported for actigraphy based devices (Zaffaroni et al., 2019).

Sleep measurement is achieved via a smartphone app, which have become ubiquitous in the last decade, eliminating the initial barrier to adoption represented by the cost and effort associated with purchasing a custom piece of hardware. The average emitted acoustic power is less than 75dB, well within the most stringent guidelines on sound exposure and the frequencies employed are above 18 KHz, above the audibility range of the vast majority of the adult population. The app utilizes a patented sensing technology and custom algorithms. Sleep monitoring can be achieved by placing a smartphone onto the bedside locker and starting the app. The app employs sophisticated algorithms to identify sleep stages: Wake (W), Light Sleep (N1, N2 sleep), Deep Sleep (N3 sleep), REM or Absence. The algorithms for the app technology were developed by using several hundred-night recordings from multiple subjects in their home consisting of concurrent measurements performed via a smartphone equipped with the Drive app and a ResMed S+ device respectively.

#### 9.4.9 Intervention and Control

The Dein Schlaf. Dein Tag. App powered by SleepScore is a personalized and dynamic digital sleep improvement program offered via smartphone. The app begins with a brief

onboarding and registration process that informs the personalized sleep advice, followed by sleep improvement personalization goals including the following potential options: sleep longer, wake up less, fall asleep easier, sharpen my mind, recharge my body, stay asleep until morning, or perfect my sleep (improve SleepScore). Users are then asked to select health-related measures that are most important for them, the regularity of their bedtime, how often they exercise, common sleep disturbances, and overall self-reported sleep quality.

Based on the user's onboarding data and nightly objective sleep tracking data, the Dein Schlaf. Dein Tag. application powered by SleepScore provides personalized evidenced-based sleep advice and sleep education content founded in the principles of sleep hygiene and cognitive behavioural skills. Additional sleep improvement features embedded within the app include weekly sleep challenges, sleep sanctuary bedroom checks, sleep sounds, smart alarm, bedtime reminders, and sleep education blogs.

To increase user engagement and adherence to tracking and sleep improvement features, the application integrates contextual reinforcement strategies through daily and weekly prompts to encourage positive sleep health-related behaviours. These prompts include smartphone push notifications, in-app overlays, and emails providing sleep education content, sleep tips, individual sleep feedback, tracking/daily log reminders.

The app uses several behaviour change techniques to improve sleep-wake functioning, including the following:

**Goal setting and planning.** Goal setting is a key component to app onboarding and the advice engine. Users can select any of the following goals: sleep longer, wake up less, fall asleep easier, sharpen my mind, recharge my body, stay asleep until morning, or perfect my sleep (improve SleepScore). Users are then asked to select health-related measures that are most important for them, the regularity of their bedtime, how often they exercise, common sleep disturbances, and overall self-reported sleep quality. The app then uses criteria to give feedback to users when they are nearing or meeting sleep improvement criteria based on these goals.

**Feedback and monitoring.** The sleep history page shows retrospective SleepScore's in order to reduce false beliefs about sleep by providing objective sleep data. In relation to goals and planning, feedback on behaviour is provided based on the measurement of objective sleep and daytime behaviours logged in the log-your-day feature.

**Shaping knowledge.** We use advice and insights based on the sleep guide and log your day items with instructions on how to remove or reduce aversive stimuli (e.g., excessive caffeine intake, excessive pre-bed light, alcohol consumption, sedentary behavior) and improve stimulus control (e.g., only using bed for sleep and intimacy).

**Natural consequences.** Information about health consequences and the salience of insufficient or poor quality sleep are provided to users in the sleep guide and research articles summarized as blog posts.

#### 9.4.10 Inclusion of users and baseline parameters

The investigator will inform eligible users about the study and the use of data. If the user is willing to participate, the informed consent form for data use will be handed out for signature. After signing by user and investigator, study relevant data will be reported after the participants has completed relevant questionnaires (see Annex1)

9.4.11 Assessments Table

| Assessment | Baseline | 6 weeks | 12 weeks |
|---|---|---|---|
| Inclusion and exclusion criteria | X | | |
| Demographics | Х | | |
| History | Х | | |
| Social status | Х | | |
| Self-report questionnaires (see Annex 1) | Х | X | Х |
| Assessment of objective sleep parameters via Dein Schlaf. Dein Tag App (each night) | Х | Х | Х |

#### 9.5 Data sources

#### 9.5.1 Data obtained from users

Baseline and 6-weeks and 12-weeks data regarding sleep, stress, and mental health questionnaires including:

| 1 | Regensburg Insomnia Scale |
|---|---------------------------------------------------|
| 2 | Schlaffragebogen B |
| 3 | Short Form 12 Health Survey Questionnaire (SF-12) |
| 4 | Pittsburgh Sleepiness Quality Index (PSQI) |
| 5 | Perceived Stress Scale (PSS) |

# 9.5.2 <u>Data imported from the Dein Schlaf. Dein Tag. App</u>

Digital data objectively measured using the Dein Schlaf. Dein Tag. App will contain the following parameters,

- Sleep stage and sleep-wake data included by not limited to total sleep time, sleep onset latency, wake after sleep onset, sleep efficiency and usage patterns.

#### 9.6 Study size

An a priori power analysis was performed using GPower version 3.1.9.7. Previous research indicates that effect sizes between 0.20 and 0.50 can be expected using a digital sleep application. A conservative approach (assuming an effect size of 0.20) will require 150 participants in each group (N=150) to detect significant effects between app group and wait-list control group for both primary and secondary outcome measures (alpha: 0.05, power: 0.80, allocation ratio 1:1). As trials with solely online recruitment may have higher drop out rates, we increased the participants in each group to 300 (total: 600 participants).

#### 9.7 Data management

Applicable national and international legal requirements for data handling and data archiving will be met. Participant study materials including recruitment materials, participant informed consent documents (PICF), study withdrawal forms, and study progress will be collected using an EU data center of Forsta/Decipher which is GDPR compliant, ISO 27001 certified, with SOC2 accredited data centers.

Objective sleep data will be collected using the Dein Schlaf. Dein Tag. application, and stored within an EU data center of the Microsoft Azure cloud system, an ISO 27001 certified and SOC 1, SOC 2, and GDPR compliant cloud service provider. Self-reported questionnaire data will be captured using an EU data center of Forsta/Decipher which is GDPR compliant, ISO 27001 certified, with SOC2 accredited data centers. Objective sleep data is encrypted in transit and at rest and additionally, personally identifiable information is hashed before being stored in the database. Access to databases for data analysis which include person identifiable information is limited to approved administration staff and is locked to the corporate IP address in the EU.

Personal information identifiers are separated from measurements so that employees of SleepScore Labs International LTD can work with accordance of least privilege to perform adequate work duties. Authentication controls are also implemented to protect customer data using passwords and usernames – external parties do not have any authentication services. Upon completion of data collection, de-identified objective data from Microsoft Azure cloud system and self-reported Forsta/Decipher data will be merged into a GDPR compliant data repository. Azure Data Factory will be used to combine the data, with processed data being stored in a Microsoft Azure SQL Server hosted in the EU. Access to this repository, which is required for analysis, will be limited to specific EU-based employees.

#### 9.7.1 Personal data and data protection

Data collected in the course of this study are subject to strict data protection measures. Objective data in the system is encrypted and secure while in transit and at rest using the latest security protocols. The data protection notice informs end-users about their data protection rights and how to exercise them (i.e. make data subject rights requests). We will comply with the requirements of Articles 12 to 21 GDPR, as applicable. All study participant data that is recorded will be pseudonymized for storage and analysis: Objective sleep data from the app as collected and controlled by SleepScore Labs and self-reported questionnaire data as collected by a vendor on behalf of ResMed Objective sleep data from the Dein Schlaf. Dein Tag. App as specified in this protocol, and without personal identifiers will be send to vendor, combined with self-reported questionnaire data by vendor and equipped with new identifiers to result in a de-identified set of study data. At the end of the project, the data will be deleted from the vendor's servers, transferred to ResMed and shared with Sleepscore Labs for joint analysis. De-identified study data will be stored at ResMed for 10 years.. Data will be collected and processed to reach the goals of the study and furthermore possible evaluations for sleep research and publications. Participants will be informed about their rights in terms of data usage, data storage, correction of data and deletion of stored data through the data protection notice. This notice sets out the data protection rights of the user and how they can exercise their data protection rights under GDPR.

#### 9.8 Data analysis

Demographic and other key study variables will be compared between intervention group and control group at the baseline using t tests for continuous variables and chi squared for categorical variables to test whether the randomization has worked adequately. The primary analysis will include all randomized participants. Secondary analyses will be conducted using an adherent to treatment approach, excluding participants who did not sufficiently engage with app throughout the study (<3 tracked nights of sleep per week, respectively used the app modules regularly).

The questionnaire data will be analyzed by an ANOVA, with one factor (app condition vs. waitlist control group) and time (Baseline, 6-weeks, 12-weeks). To handle missing values, a mixed-model approach with the same factors will be applied. The critical statistical test would be the interaction term between app condition and the waitlist control group.

For objectively recorded sleep data, repeated measured data will be analyzed using multi-level modeling (MLM) in a nested way (nights within participants), will be performed allowing for analyzing changes with the intervention (app) group. To evaluate changes in primary and secondary outcome measures assessed by validated scales at baseline, 6-weeks, and 12-weeks, we will compare within-group differences for each time-point using a t-test if normally distributed, or the Mann Whitney-U test for non-normally distributed continuous data. In addition, effect sizes for the changes within both groups (questionnaire data) and app group (objective sleep parameters) will be computed.

#### 9.9 Quality control

Quality control is defined as the operational techniques and activities, such as monitoring, undertaken within the quality assurance system to verify that the requirements for quality of the study related activities have been fulfilled. Quality control should be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Quality assurance is defined as the planned and systematic actions that are established to ensure that the study is performed, and the data generated, documented (recorded) and reported, in compliance with Good Clinical Practice (GCP) and the applicable regulatory requirements.

#### 9.9.1 Access to Source Data/Document

The investigator will permit, and participating subjects will consent for, potential study-related monitoring, audits, Ethics Committee review and regulatory inspections, providing direct access to primary participant's data (i.e. source data) that support data in the Microsoft Azure cloud. Direct access is defined as the permission to examine, analyze, verify and reproduce any records and reports that are important to evaluation of a study. Any party (e.g. domestic and foreign regulatory authorities, the sponsor and/or authorized representatives of the sponsor such as monitors and auditors) with direct access should take all reasonable precautions within the constraints of the applicable regulatory requirements to maintain the confidentiality of users identities and sponsor proprietary information.

#### 9.9.2 Quality assurance:

Quality assurance is defined as the planned and systematic actions that are established to ensure that the study is performed, and the data are generated, documented (recorded) and reported in compliance with GCP and the applicable regulatory requirements.

#### 9.10 Study monitoring

The sponsor or authorized, qualified representatives of the sponsor will accomplish the monitoring during the study. Source documents will be reviewed for verification of consistency. The investigator agrees that representatives or the designees of the sponsor, and appropriate regulatory bodies will be given direct access to the regular files of the user. It is important that the investigator and their relevant personnel are available during the monitoring visits and possible audits and that an appropriate location and sufficient amount of time is devoted to the process. During the monitoring visit a PC with internet connection should be available to the monitor for direct connection to the internet database of the study and to all the data of the users if stored in the data system.

#### 9.10.1 Audit

An audit is a systematic and independent review of study related activities and documents to determine whether the validated study related activities were conducted and the data were recorded, analyzed and accurately reported according to the protocol, designated Standard Operating Procedure (SOPs), GCP and the applicable regulatory requirements.

#### 9.11 Limitations of the research methods

It is expected that variations in the use of the Dein Schlaf. Dein Tag will occur, i.e., some users will use the app very intensely, others might use it regularly but not so intense. Due to the expected of variations in procedures and in particular in usage times of the sleep advice engine, the magnitude of statistical significance (i.e., effect size) is expected to be smaller but still within the range of 0.20 to 0.50.

#### 9.12 Other aspects

None

#### 10. Protection of human subjects

All sleep advice engine support activities used are decided individually by the user and are not pre-defined by the study protocol. All sleep advice engine support activities are to be used in line with their marketing authorisation. Participation does not pose additional risks and adverse events are not expected given the behavioural nature of the intervention. All Sleep advice engine support activities are performed in accordance with all applicable ethical and regulatory standards. Before initiating the study in a country, approval of the IRB / IEC will be obtained.

#### 11. Management and reporting of Adverse Events/Adverse Reactions

Unanticipated problems or any unexpected adverse events will be promptly reported by the PI to an IRB representative from the Ethik-Kommission der Medizinischen Fakultät der Universität Duisburg-Essen by phone (+49 (0) 201 - 723 3448) or email (ethikkommission@uk-essen.de), as well as any other medium (e.g. faxed form) requested by the 3rd party IRB following email/phone notification.

#### 12. Plans for disseminating and communicating study results

Study results will be pooled for the purpose of publication that will be jointly coordinated by SleepScore Labs and ResMed. Preparation of the comprehensive publication will occur at the completion of the study. Publications arising from this study will be jointly defined, executed, and published or alternately consented by both sides.

| | _ | |
|------------|---|-----------------|
| Annex 1. ( | 1 | IIIDETIANNAIRDE |
| Alliex I. | , | uestionnaires |

| | Items | Recruitment | Baseline | 6<br>Weeks | 12<br>Weeks | Purpose |
|---|---|---|---|---|---|---|
| Regensburg<br>Insomnia Scale | 10 | Х | | | | Eligibility |
| SF-B | 29 | | X | X | X | Effect on sleep |
| SF-12 | 12 | | X | X | X | Effect on preventative health |
| Pittsburgh Sleep<br>Quality Index<br>(PSQI) | 19 | | X | Х | X | Effect on sleep quality |
| Perceived<br>Stress Scale | 10 | | Х | Х | Х | Effect on<br>Stress |

#### Annex 2. References

Dein Schlaf. Dein Tag. App: Zaffaroni A., Coffrey S., Dodd S., Kilron H., Lyon G., O'Rourke D., Lederer K., Fietze I., Penzel T. Sleep stage monitoring based on sonar smartphone technology. Annu Int Conf IEEE Eng Med Biol Soc. 2019; 2019:2230-2233.

LISST: Landecker Inventar zur Erfassung von Schlafstörungen; Hans-Günter Weeß, Enzyklopädie der Schlafmedizin, 2020, 1-2; DOI: 10.1007/978-3-642-54672-3 261-1

Munich Chronotype Questionnaire: Ghotbi, N., Pilz, L. K., Winnebeck, E. C., Vetter, C., Zerbini, G., Lenssen, D., Frighetto, G., Salamanca, M., Costa, R., Montagnese, S., & Roenneberg, T. (2019). The μMCTQ: An Ultra-Short Version of the Munich ChronoType Questionnaire. Journal of Biological Rhythms, 1, 98–110.

Perceived Stress Scale: Klein, E. M., Brähler, E., Dreier, M., Reinecke, L., Müller, K. W., Schmutzer, G., Wölfling, K., & Beutel, M. E. (2016). The German version of the Perceived Stress Scale – psychometric characteristics in a representative German community sample. BMC Psychiatry, 1.

PSQI: Backhaus, J., Junghanns, K., Broocks, A., Riemann, D., & Hohagen, F. (2002). Test–retest reliability and validity of the Pittsburgh Sleep Quality Index in primary insomnia. Journal of Psychosomatic Research, 3, 737–740.

Regensburg Insomnia Scale: Crönlein, T., Langguth, B., Popp, R., Lukesch, H., Pieh, C., Hajak, G., & Geisler, P. (2013). Regensburg Insomnia Scale (RIS): a new short rating scale for the assessment of psychological symptoms and sleep in insomnia; Study design: development and validation of a new short self-rating scale in a sample of 218 patients suffering from insomnia and 94 healthy controls. Health and Quality of Life Outcomes, 1, 65.

SF-12: Standardization of the SF-12 Version 2.0 Assessing Health-Related Quality of Life in a Representative German Sample; Wirtz, Markus Antonius; Morfeld, Matthias; Glaesmer, Heide; Brähler, Elmar; Diagnostica, 2018, Vol 64 (4), 215-226

SF-B: Schredl, M., Schenck, W., Görtelmeyer, R. *et al.* Einflußfaktoren auf die Schlafqualität bei Gesunden. *Somnologie* 2, 99–103 (1998).

#### **Certificate Of Completion**

Envelope Id: 2E1EED059FEE428FA7ECB252516D767C

Subject: Complete with DocuSign: SleepScoreLabs\_Resmed Project\_Protocol\_V28Apr2023\_.pdf

Source Envelope:

Document Pages: 23 Signatures: 3 Certificate Pages: 5 Initials: 0

AutoNav: Enabled

**Envelopeld Stamping: Enabled** 

Time Zone: (UTC+01:00) Amsterdam, Berlin, Bern, Rome, Stockholm, Vienna

Status: Sent

**Envelope Originator:** Oliver.Munt@ResMed.de 125 Technology Pkwy

Peachtree Corners, GA 30092 Oliver.Munt@ResMed.de IP Address: 163.116.173.57

#### **Record Tracking**

Status: Original Holder: Oliver.Munt@ResMed.de Location: DocuSign

DocuSigned by:

04FB954265AE4BF...

Daniela Ehrsam-Tosi

Signature Adoption: Pre-selected Style Using IP Address: 163.116.175.20

Signature Adoption: Pre-selected Style Using IP Address: 76.32.114.7

Oliver.Munt@ResMed.de

Sent: 5/5/2023 9:13:03 AM

Sent: 5/5/2023 9:13:01 AM

Viewed: 5/7/2023 6:23:44 PM

Signed: 5/7/2023 6:23:58 PM

Sent: 5/5/2023 9:13:02 AM

Viewed: 5/7/2023 1:34:03 AM

Signed: 5/9/2023 5:26:24 PM

Sent: 5/5/2023 9:13:03 AM

Viewed: 5/8/2023 8:53:56 AM

Signed: 5/8/2023 8:54:49 AM

**Timestamp** 

### Signer Events Christoph Schöbel

Signature

Christoph.Schoebel-Extern@ResMed.de Security Level: Email, Account Authentication

(None)

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

5/5/2023 9:07:55 AM

Daniela Fhrsam-Tosi

(None)

Daniela.Ehrsam-Tosi@resmed.ch Security Level: Email, Account Authentication

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

Elie.Gottlieb@sleepscorelabs.com

Security Level: Email, Account Authentication

(None)

Elie Gottlieb

**Electronic Record and Signature Disclosure:** 

Accepted: 5/7/2023 1:34:03 AM

ID: 3e8cff50-3f80-451a-9fc0-3c1b95c8d9fb

Susanne Fischer

Susanne.Fischer@resmed.de

Security Level: Email, Account Authentication

(None)

DocuSigned by:

Plie Gottlieb

A7169A2AE3DD47E..

Signed using mobile

Susanne Fischer

Signature Adoption: Pre-selected Style

B6337AFF84D74C4...

Using IP Address: 163.116.173.75

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|-------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |

| Intermediary Delivery Events | Status | Timestamp |
|---|---|---|
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 5/5/2023 9:13:04 AM |
| Certified Delivered | Security Checked | 5/8/2023 8:53:56 AM |
| Signing Complete | Security Checked | 5/8/2023 8:54:49 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, ResMed Ltd (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact ResMed Ltd:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: andrew.hunter@resmed.com.au

#### To advise ResMed Ltd of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at andrew.hunter@resmed.com.au and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

## To request paper copies from ResMed Ltd

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to andrew.hunter@resmed.com.au and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with ResMed Ltd

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to andrew.hunter@resmed.com.au and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|----------------------------|----------------------------------------------|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | |
| | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy |
| | Server must enable HTTP 1.1 settings via |
| | proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify ResMed Ltd as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by ResMed Ltd during the course of my relationship with you.